CLINICAL TRIAL: NCT00670709
Title: Examination of Quantitative Electroencephalographic Biomarkers in Huntington's Disease: A Pilot Project
Brief Title: Examination of Quantitative Electroencephalographic (QEEG) Biomarkers in Huntington's Disease
Acronym: HD
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: High Q Foundation (Unknown)
Responsible Party: Principal Investigator, Andrew F. Leuchter, Andrew F. Leuchter, M.D., University of California, Los Angeles
Other Study IDs: QEEG and HD
Record Dates: First submitted 2008-04-30; First posted 2008-05-02 (Estimated); Results first posted 2010-08-16 (Estimated); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Huntington's Disease
Keywords: encephalography; quantitative; biomarkers
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Subjects with mild or moderate Huntington's Disease
- 2: Normal Controls

SUMMARY:
The pace of basic science research defining the mechanisms of selective neuronal degeneration in Huntington disease (HD) has far exceeded the pace of translation of this information into clinically effective treatments for the disease. One reason for this bottleneck between bench and bedside is the paucity of available surrogate markers for HD. Identification of surrogate markers is critical for the design of future clinical trials. Such markers could provide a reliable signal of early brain dysfunction in HD and could be used as a biomarker in trials of agents that could prevent onset or delay progression of disease.

Frontal-subcortical networks are known to be affected in HD and contribute to the cognitive dysfunction characteristic of the disease. Quantitative EEG (QEEG) can be used to assess the integrity of this circuitry; characteristic QEEG abnormalities long have been known to be present in the early stages of the illness (Bylsma et al., 1994). More recent research has suggested that a comprehensive topographic approach to QEEG analysis may reveal additional changes in brain activity (Bellotti et al., 2004) that may be indicative of subclinical disease (de Tommaso et al., 2003). This proposal aims to determine whether quantitative EEG techniques can be used to identify HD-specific abnormalities and thus serve as surrogate markers of disease.

The goals of this pilot project are three-fold. First, we will determine if there are QEEG differences between normal control subjects and those with mild or moderate HD. Second, we will examine associations between severity of HD and the QEEG differences detected and determine if these QEEG differences are present when comparing the least affected HD subjects and normal controls. Third, we will examine associations between QEEG variables of interest and other clinical variables, including age of onset of symptoms, number of CAG repeats, severity of motor and behavioral symptoms as measured by the Unified Huntington Disease Rating Scale (UHDRS) subscores, and severity of cognitive impairment as measured by the cognitive subscore of the UHDRS and Mini-Mental State Examination (MMSE).

DETAILED DESCRIPTION:
We will examine three subject groups in this study: those with mild HD, those with moderate HD, and normal controls. Fifteen subjects will be examined in each group, for an overall total of forty-five subjects. HD subjects will be recruited from the UCLA Huntington Disease Center of Excellence where they have been followed with serial neurologic examinations and completion of all portions of the UHDRS every 6-12 months. Subjects that have been given a diagnosis of HD based on appropriate motor signs and a confirmatory genetic test or a known family history of HD will be invited to participate. Healthy control subjects will be recruited from the clinic as well through spouses or other unaffected relatives of patients. In addition, control subject data acquired from previous studies will be used after matching for age. All subjects will be over the age of 21 and free of other medical illnesses that could also affect brain function and will be able to give informed consent. Mild HD is defined as having Total Functional Capacity [TFC] scores on the UHDRS of 11-13, moderate is defined as TFC of 7-10, and normal control subjects will be free of any neurologic or psychiatric illness. Subjects will be free of antipsychotic or antidepressant medications, benzodiazepines, or other medications known to affect central nervous system function for at least 10 days prior to QEEG examination.

All subjects will undergo QEEG recording in a manner similar to that employed clinically, using procedures that have been approved in other protocols by the UCLA Medical IRB and that are consistent with standard clinical EEG procedures promulgated by ABRET (American Board of Registered Electroencephalographic Technologists). Recording electrodes are applied to the scalp using an electrode cap (ElectroCap, Inc., Eaton OH); electrodes are arrayed to record electrical activity from all major brain regions using a standard extension of the International 10-20 system (figure 1). Recording electrodes are connected to an isolation amplifier that is part of the digital EEG system (NuAmp System, NeuroScan, Inc., El Paso, TX). Data are recorded in real-time on computer disk. During recording, subjects will be resting in a quiet room with subdued lighting, in the eyes-closed, maximally alert state; the EEG technologists will alert the subjects whenever drowsiness is evident on the computer monitor. Data will be displayed in real-time on a computer monitor during recording, with adjustable filtering and amplification to facilitate identification of EEG patterns as well as artifact. Data will be collected using a bandpass filter of 0.3 to 70 Hz, and will be digitized at a rate of 250 samples/channel/second. Data will be recorded with a Pz referential montage, and the NeuroScan software then will reformat the data into bipolar montages as needed for the cordance calculations. Three EOG leads will be used (RIO-A2, ROC-A2, and LOC-A1) so that lateral, horizontal, or oblique eye movement artifact may be detected easily. Data for quantitative analysis will be selected from the data recorded according to standard procedures: each EEG will be reviewed by a technician and the first 20-32 seconds of artifact-free data will be selected to be processed to obtain absolute and relative power in four frequency bands (0.5-4 Hz, 4-8 Hz, 8-12 Hz, and 12-20 Hz) after the selections are confirmed by a second technician; both technicians will be blinded to clinical status while making or reviewing the selections.

Two QEEG measures will be calculated for each subject. The first of these is cordance, which will be calculated using an algorithm that has been detailed elsewhere (Leuchter et al., 1999). Cordance is based upon a normalization of absolute and relative power values across all electrode sites and all frequency bands for a given recording. Cordance values have a stronger association with cerebral perfusion in brain tissue underlying each electrode site than do standard QEEG power measures. The second QEEG measure to be examined is QEEG coherence (Leuchter et al., 1992; 1994b), a measure of the shared functional activity between brain regions. Coherence values range between 0 - 1 and are analogous to a correlation coefficient, with values near 1 signifying highly coordinated cerebral activity. Coherence reflects not only cortical activity, but also the function of deep gray matter structures that coordinate cortical activity as well as white-matter tracts connecting brain regions.

ELIGIBILITY:
Inclusion criteria:

* Subjects affected by HD or those who are at risk for HD by virtue of having a first-degree relative with the illness, methamphetamine abuse or dependence, as well as normal controls, can participate.
* All subjects will be above the age of 21.
* Subjects will be recruited from clinical settings, and will also be self-referred.

Exclusion criteria:

* Individuals with pacemakers, infusion pumps, or metallic shrapnel will be excluded from MRI assessments.
* Such implanted metals may be attracted by the MRI machine and put the individual at risk.
* Moreover, individuals with a history of brain surgery and/or skull fracture will also be excluded.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 subjects with mild or moderate Huntington's Disease and 15 healthy normal controls
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2006-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew F Leuchter, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Laboratory of Brain, Behavior,a nd PHarmacology, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began September 2006 and ended in February 2008. All recruitment took place at UCLA Neurology Clinic and the UCLA Semel Institute.
Groups:
- Huntington Disease: Subjects with mild or moderate Huntington's Disease
- Healthy Controls: Healthy control subjects
Period: Overall Study
Arm/Group | Huntington Disease | Healthy Controls
Started | 27 | 15
Completed | 27 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Huntington Disease | Healthy Controls | Total
Number analyzed (Participants) | 27 | 15 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 15 | 42
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (11.3) | 47.3 (9.7) | 46.85 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 16 | 7 | 23
Region of Enrollment [Number; unit: participants]
  United States | 27 | 15 | 42

OUTCOME MEASURES:

1. Primary Outcome: Quantitative Electroencephalography Absolute Delta Power.
Description: Absolute power in the delta frequency as measured by quantitative electroencephalography
Time Frame: baseline- one time point
Measure: Mean (Standard Deviation); unit: microvolts squared
Arm/Group | Huntington Disease | Healthy Controls
Number analyzed (Participants) | 27 | 15
microvolts squared | 43.45 (10.83) | 10.11 (3.01)
Statistical Analysis 1: Comparison: Huntington Disease vs Healthy Controls; Test type: Superiority or Other; p < 0.0000001, t-test, 2 sided

2. Primary Outcome: Quantitative Electroencephalography Absolute Alpha Power.
Description: Absolute power in the alpha frequency as measured by quantitative electroencephalography
Time Frame: baseline EEG
Measure: Mean (Standard Deviation); unit: microvolts squared
Arm/Group | Huntington Disease | Healthy Controls
Number analyzed (Participants) | 27 | 15
microvolts squared | 56.09 (62.61) | 18.12 (15.04)
Statistical Analysis 1: Comparison: Huntington Disease vs Healthy Controls; HD subjects vs control subjects; Test type: Superiority or Other; p < 0.005, t-test, 2 sided

ADVERSE EVENTS:
Description: There reason there was no serious adverse events and no other adverse events listed is because this was not a treatment study. It was an observed study, with no patients treated during the process. Therefore, there were no serious adverse events and no other adverse events recorded.
Arm/Group | Huntington Disease | Healthy Controls
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No